CLINICAL TRIAL: NCT02025894
Title: Risk Factors for Thromboembolic and Infectious Complications Related to Percutaneous Central Venous Catheters in Cancer - Prospective Multicenter Study
Acronym: ONCOCIP
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-01; 2010-A01064-35 (Other: French ministry of health)
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2013-12

CONDITIONS: Cancer
Keywords: neoplastic solid tumour; PCVC; thromboembolic complications; infectious complications; risk factors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCVCs: Cohort of cancer patients with indication PCVC under the usual practice

SUMMARY:
The purpose of this study is to identify risk factors for thromboembolic and /or infectious complications in 3,000 patients with solid tumor and receiving a Percutaneous Central Venous Catheter (PCVC). A better understanding of the risk factors for these complications in this population would then allow interventional studies to be proposed to assess the benefit of prophylactic procedures in a sub-group of patients at most risk.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a neoplastic solid tumour with an indication for insertion of a PCVC.

Exclusion Criteria:

* Haematological neoplasm pathology, PCVC removal scheduled within 2 weeks of insertion,
* Therapeutic doses of anticoagulants required at inclusion,
* PCVC inserted by the femoral vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of consecutive patients
Sampling Method: Non-Probability Sample
Enrollment: 3032 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Thromboembolic complications: | one year
Locoregional or disseminated infectious complications: | one year

SECONDARY OUTCOMES:
Medical and economic consequences of these complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fournel, MD, Principal Investigator — Institut Cancérologique Lucien Neuwirth; Hervé DECOUSUS, MDPhD, Study Director — CIC - CHU DE SAINT-ETIENNE; Franck CHAUVIN, MDPhD, Study Director — Institut cancérologique Lucien Neuwirth
Locations (27):
- France (27):
  - CH d'Annecy, Annecy, France
  - CH Intercommunal Annemasse-Bonneville, Annemasse, France
  - Polyclinique de Savoie, Annemasse, France
  - CH Chambéry, Chambéry, France
  - CHU Clermont-Ferrand, Clermont-Ferrand, France
  - Pôle Santé république, Clermont-Ferrand, France
  - CH Feurs, Feurs, France
  - Institut Daniel Hollard, Grenoble, France
  - CH EmileRoux, Le Puy-en-Velay, France
  - CH Lyon Sud, Lyon, France
  - Clinique de la sauvergarde, Lyon, France
  - Clinique Eugène André, Lyon, France
  - Clinique Portes du Sud, Lyon, France
  - Clinique Saint-Joseph Saint-Luc, Lyon, France
  - Hôpital de la Croix Rousse, Lyon, France
  - Hôpital Desgenettes, Lyon, France
  - Hôpital privé Jean-Mermoz, Lyon, France
  - Infirmerie Protestante, Lyon, France
  - CH de Montbrison, Montbrison, France
  - CH de Roanne, Roanne, France
  - CH Pays du Gier, Saint-Chamond, France
  - CHU Saint-Etienne Service de Gynécologie, Saint-Etienne, France
  - CHU Saint-Etienne Service de Gastroentérologie, Saint-Etienne, France
  - Hôpital privé de la Loire, Saint-Etienne, France
  - Institut Cancérologique Lucien neuwirth, Saint-Priest-en-Jarez, France
  - Hôpitaux du Léman, Thonon-les-Bains, France
  - Hôpital Privé Drôme Ardèche, Valence, France

REFERENCES:
- [Background] Agnelli G, George DJ, Kakkar AK, Fisher W, Lassen MR, Mismetti P, Mouret P, Chaudhari U, Lawson F, Turpie AG; SAVE-ONCO Investigators. Semuloparin for thromboprophylaxis in patients receiving chemotherapy for cancer. N Engl J Med. 2012 Feb 16;366(7):601-9. doi: 10.1056/NEJMoa1108898. PMID 22335737
- [Background] Debourdeau P, Farge D, Beckers M, Baglin C, Bauersachs RM, Brenner B, Brilhante D, Falanga A, Gerotzafias GT, Haim N, Kakkar AK, Khorana AA, Lecumberri R, Mandala M, Marty M, Monreal M, Mousa SA, Noble S, Pabinger I, Prandoni P, Prins MH, Qari MH, Streiff MB, Syrigos K, Buller HR, Bounameaux H. International clinical practice guidelines for the treatment and prophylaxis of thrombosis associated with central venous catheters in patients with cancer. J Thromb Haemost. 2013 Jan;11(1):71-80. doi: 10.1111/jth.12071. PMID 23217208
- [Background] Saber W, Moua T, Williams EC, Verso M, Agnelli G, Couban S, Young A, De Cicco M, Biffi R, van Rooden CJ, Huisman MV, Fagnani D, Cimminiello C, Moia M, Magagnoli M, Povoski SP, Malak SF, Lee AY. Risk factors for catheter-related thrombosis (CRT) in cancer patients: a patient-level data (IPD) meta-analysis of clinical trials and prospective studies. J Thromb Haemost. 2011 Feb;9(2):312-9. doi: 10.1111/j.1538-7836.2010.04126.x. PMID 21040443
- [Background] Akl EA, Kamath G, Yosuico V, Kim SY, Barba M, Sperati F, Cook DJ, Schunemann HJ. Thromboprophylaxis for patients with cancer and central venous catheters: a systematic review and a meta-analysis. Cancer. 2008 Jun;112(11):2483-92. doi: 10.1002/cncr.23479. PMID 18404702
- [Background] Mollee P, Jones M, Stackelroth J, van Kuilenburg R, Joubert W, Faoagali J, Looke D, Harper J, Clements A. Catheter-associated bloodstream infection incidence and risk factors in adults with cancer: a prospective cohort study. J Hosp Infect. 2011 May;78(1):26-30. doi: 10.1016/j.jhin.2011.01.018. Epub 2011 Apr 2. PMID 21459476
- [Background] Chaukiyal P, Nautiyal A, Radhakrishnan S, Singh S, Navaneethan SD. Thromboprophylaxis in cancer patients with central venous catheters. A systematic review and meta-analysis. Thromb Haemost. 2008 Jan;99(1):38-43. doi: 10.1160/TH07-07-0446. PMID 18217132
- [Background] Khorana AA, Francis CW, Blumberg N, Culakova E, Refaai MA, Lyman GH. Blood transfusions, thrombosis, and mortality in hospitalized patients with cancer. Arch Intern Med. 2008 Nov 24;168(21):2377-81. doi: 10.1001/archinte.168.21.2377. PMID 19029504
- [Background] Schwarz RE, Groeger JS, Coit DG. Subcutaneously implanted central venous access devices in cancer patients: a prospective analysis. Cancer. 1997 Apr 15;79(8):1635-40. PMID 9118051
- [Derived] Decousus H, Bourmaud A, Fournel P, Bertoletti L, Labruyere C, Presles E, Merah A, Laporte S, Stefani L, Piano FD, Jacquin JP, Meyer G, Chauvin F; ONCOCIP Investigators. Cancer-associated thrombosis in patients with implanted ports: a prospective multicenter French cohort study (ONCOCIP). Blood. 2018 Aug 16;132(7):707-716. doi: 10.1182/blood-2018-03-837153. Epub 2018 Jul 6. PMID 29980524